CLINICAL TRIAL: NCT02249169
Title: Developing Novel Microbiota-Targeted Therapies for Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, PI, Mayo Clinic
Other Study IDs: 14-000305
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, whole blood, stool, colonic mucosal tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- IBS-C: Patients with a clinical diagnosis of constipation-predominant irritable bowel syndrome
- IBS-D: Patients with a clinical diagnosis of diarrhea-predominant irritable bowel syndrome
- Healthy subjects: Subjects without a clinical diagnosis of IBS-C or IBS-D
- Healthy Controls: Subject without a clinical diagnosis of IBS-C or IBS-D and who is either a first-degree relative of an IBS participant or is not genetically related but resides with the IBS participant

SUMMARY:
This longitudinal study is being done to understand mechanisms underlying development of irritable bowel syndrome (IBS) and the role of the gut bacteria in development of symptoms. This information will be used to determine whether temporal changes in gut microbial taxonomy and metabolism are associated with changes in symptom severity in IBS, and if targeted dietary interventions, including prebiotics, can reverse or moderate these changes.

ELIGIBILITY:
IBS-C and IBS-D SUBJECTS:

Inclusion Criteria:

* Clinical diagnosis of IBS-C or IBS-D
* Age 18 to 65

Exclusion Criteria:

* Prior history of abdominal surgeries (except appendectomy and cholecystectomy)
* Known diagnosis of inflammatory bowel disease, microscopic colitis, celiac disease or other inflammatory condition
* Antibiotic use within the past 4 weeks (they can be enrolled after a four-week washout period and subsequent use during the 6-month study duration does not exclude them)
* Bleeding risk or medications which may increase risk of bleeding for patients who agree to undergo flexible sigmoidoscopy
* Bowel preparation for colonoscopy within the past week
* Pregnancy or plans to become pregnant within the study time frame
* Vulnerable adults
* Age greater than or equal to 66
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of the study, would increase risks of flexible sigmoidoscopy (for those opting for this), or in the judgment of the investigator would potentially interfere compliance to this study or would adversely affect study outcomes

HEALTHY SUBJECTS:

Inclusion Criteria:

* Age 18 to 65
* No clinical diagnosis of IBS-C or IBS-D

Exclusion Criteria:

* Prior history of abdominal surgeries (except appendectomy and cholecystectomy)
* Known diagnosis of inflammatory bowel disease, microscopic colitis, celiac disease or other inflammatory condition
* Antibiotic use within the past 4 weeks (they can be enrolled after a four-week washout period and subsequent use during the 6-month study duration does not exclude them)
* Bleeding risk or medications which may increase risk of bleeding for patients who agree to undergo flexible sigmoidoscopy
* Bowel preparation for colonoscopy within the past week
* Pregnancy or plans to become pregnant within the study time frame
* Vulnerable adults
* Age greater than or equal to 66
* Any other disease(s), condition(s) or habit(s) that would interfere with completion of the study, would increase risks of flexible sigmoidoscopy (for those opting for this), or in the judgment of the investigator would potentially interfere compliance to this study or would adversely affect study outcomes
* Clinical diagnosis of IBS-C or IBS-D

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Motility Clinic, Clinical Research Unit, GI Department
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiome in patients with IBS compared to healthy individuals measured over 6 months | baseline, 6 months
  Participants will provide a stool sample at baseline and at periodic intervals for 6 months to assess gut microbial composition.

CONTACTS AND LOCATIONS:
Overall Officials: Purna C. Kashyap, M.B.B.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials